CLINICAL TRIAL: NCT05901220
Title: Joint School-Health Project of the Neapolitan Child
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Professor, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Federico II-Cardarelli
Record Dates: First submitted 2023-05-06; First posted 2023-06-13 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: No Condition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Students of a school in the Campania region (Experimental)
  Interventions: Behavioral: Healthy lifestyle

INTERVENTIONS:
Behavioral: Healthy lifestyle — An educational programme to promote healthy lifestyle will be performed.

SUMMARY:
Unhealthy lifestyle habits during the childhood could negatively impact the health status actual and during the later stages of life.

The School represents the major Institution to implement actions aim at promoting healthy lifestyles habits.

The Joint School-Health Project of the Neapolitan Child aimed at assessing the impact of a health education programme to improve lifestyle habits during the childood. To evalute the effects of this educational programme, the dietary habits, the sleep hours, the hours spent in sedentary behaviors (tv, smartphone) and the hours of physical activity will be evaluate at the baseline and at the end of the programme.

ELIGIBILITY:
Inclusion Criteria:

* students aged 5-13 years of both sex;
* parents/tutor written informed consent.

Exclusion Criteria:

* lack of written informed consent;
* unwillingness to participate.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 223 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Intake of energy and nutrients | 7-day
  A 7-day food diary to evaluate the dietary intake of energy and nutrients.
Intake of ultraprocessed foods | 7-day
  A 7-day food diary to evaluate the dietary intake of ultraprocessed foods.
Intake of dietary advanced glycation end-products | 7-day
  A 7-day food diary to evaluate the dietary intake of the detrimental compounds of ultraprocessed foods, the advanced glycation end-products.
Adherence to the Mediterranean Diet | 9 months
  The KIDMED questionnaire is used to evaluate the adherence to the Mediterranean Diet. The total score is 12 points and a score of ≤3 means 'very low', between 4-7 'moderate' and ≥8 refers to 'high' adherence to the Mediterranean Diet
The sleep habits | 9 months
  The Italian Children's Sleep Habits Questionnaire is used to evaluate the sleep habits. The total score is the sum of the 10 responses obtained on each item and the highest scores indicate the worst sleep habits.
The hours spent in sedentary behaviors | 9 months
  The WHO-Collaborative Health Behaviour in School-aged Children (HBSC) study questionnaire is used to evaluate the hours spent in sedentary behaviors (tv, smartphone, etc). Three items assess sedentary screen-based activities: 1) "About how many hours a day do you usually watch television (including DVDs and videos) in your free time?" 2) "About how many hours a day do you usually play games on a computer or games console (Playstation, Xbox, GameCube etc.) in your free time?" and 3) "About how many hours a day do you usually use a computer for chatting on-line, internet, emailing, homework etc. in your free time? All three items have nine possible responses: "none at all", about 30 min, 1 hour, 2 hour, up to ≥7 hour/day. Responses for weekdays are recoded into ≤ versus > 2 hour/day.
The hours of physical activity | 9 months
  The WHO-Collaborative Health Behaviour in School-aged Children (HBSC) study questionnaire is used to evaluate the hours of physical activity. Moderate to vigorous physical activity (MVPA) is assessed by asking: "On how many days in the past week were you physically active for 60 minutes or more". Physical activity was defined as "any activity that increases your heart rate and makes you get out of breath some of the time" with examples of such activities. Response categories were: "0 days", "1", "2", etc up to "7 days", recoded as < or ≥ 5 times/week17. Vigorous physical activity (VPA) is assessed by asking: "Outside school hours, how many hours a week do you usually exercise in your free time so much that you get out of breath or sweat?" Response categories are none, about 30 minutes, and 1, 2-3, 4-6, ≥7 hours; recoded into < or ≥ 2 hour/week.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No